CLINICAL TRIAL: NCT03258190
Title: Lime Powder Regimen Supplement Alleviates Urinary Metabolic Abnormalities to Prevent Urolithiasis Recurrence.
Brief Title: Lime Powder Regimen (LPR) for Prevention of Renal Stone Recurrence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Sanpasitthiprasong Hospital (Other Government); Burapha University (Other)
Responsible Party: Principal Investigator, Piyaratana Tosukhowong, Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LPR0001
Record Dates: First submitted 2017-08-20; First posted 2017-08-23 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Urolithiasis
Keywords: Urolithiasis; Recurrence; Citrate; Antioxidants; Lime Powder Regimen
MeSH Terms: conditions — Urolithiasis; Recurrence

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant
Masking Description: LPR and Placebo were prepared in the same containers with code that was provided by investigators
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lime Powder Regimen (Experimental): Participants were asked to take LPR twice a day for 6 months
  Interventions: Drug: Lime Powder Regimen
- Placebo (Placebo Comparator): Participants were asked to take Placebo twice a day for 6 months
  Interventions: Drug: Lime Powder Regimen

INTERVENTIONS:
Drug: Lime Powder Regimen — LPR and placebo were randomly given to subjects for 6 months
  Other Names: LPR supplement

SUMMARY:
Lime powder regimen (LPR) is a lime-derived composition enriches with citrate/citric acid and potassium. LPR was invented to treat the renal stone patients with high risk of stone recurrence after stone removal. LPR should have equal or higher efficacy and lower adverse effect than current standard medicine.

DETAILED DESCRIPTION:
Lime powder regimen (LPR) is a mixture of lime-derive component with adjuvants containing high concentration of citrate, and moderate amount of potassium, magnesium and antioxidants. LPR was tested and verified to be very less toxic in cell culture and animal models. The clinical trial phase II showed that LPR reduced urinary metabolic abnormalities that enhance stone formation, such as hypocitraturia, hypokaliuria and acidified urine. Adverse effect of LPR was very low.

ELIGIBILITY:
Inclusion Criteria:

* Renal stone patients who were identified and stone was removed by surgical method.

Exclusion Criteria:

* Chronic kidney disease, chronic liver disease, history of coronary artery disease, or person who takes any medication that alters urinary metabolic profiles

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Renal stone recurrence | 6 months
  The stone recurrence after surgical removal of stone that can be detected by CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chariyavilaskul P, Poungpairoj P, Chaisawadi S, Boonla C, Dissayabutra T, Prapunwattana P, Tosukhowong P. In vitro anti-lithogenic activity of lime powder regimen (LPR) and the effect of LPR on urinary risk factors for kidney stone formation in healthy volunteers. Urolithiasis. 2015 Apr;43(2):125-34. doi: 10.1007/s00240-015-0751-y. Epub 2015 Jan 15. PMID 25588323
- See also: Clinical trial phase 1 — https://www-ncbi-nlm-nih-gov.cuml1.md.chula.ac.th/pubmed/?term=In+vitro+anti%E2%80%91lithogenic+activity+of+lime+powder+regimen+(LPR)+and+the+effect+of+LPR+on+urinary+risk+factors+for+kidney+stone+formation+in+healthy+volunteers